CLINICAL TRIAL: NCT04309578
Title: A Phase II Clinical Study of Trastuzumab in Combination With Capecitabine and Cisplatin (XP) in Patients With Tissue HER2-negative But Serum HER2-positive Advanced Gastric Cancer: XP+Samfenet
Brief Title: A Study of Trastuzumab in Combination With Capecitabine and Cisplatin in Patients With Tissue HER2- But Serum HER2+ AGC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2002
Record Dates: First submitted 2020-01-06; First posted 2020-03-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastric or Gastroesophageal Junction(GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Trastuzumab; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Single arm
  Interventions: Drug: Trastuzumab, Capecitabine and Cisplatin

INTERVENTIONS:
Drug: Trastuzumab, Capecitabine and Cisplatin — * Trastuzumab intravenous administration at a loading dose of 8 mg/kg on day 1 followed by 6 mg/kg every 3 weeks
  * Capecitabine oral administration at a dose of 1000 mg/m2 twice daily for 14 days every 3 weeks (from evening on day 1 to morning on day 15)
  * Cisplatin intravenous administration at a dose of 80 mg/m2 on day 1

SUMMARY:
A phase II clinical study of trastuzumab in combination with capecitabine and cisplatin (XP) in patients with tissue HER2-negative but serum HER2-positive advanced gastric cancer

DETAILED DESCRIPTION:
3-weekly/ 1cycle treatment

* Trastuzumab intravenous administration at a loading dose of 8 mg/kg on day 1 followed by 6 mg/kg every 3 weeks
* Capecitabine oral administration at a dose of 1000 mg/m2 twice daily for 14 days every 3 weeks (from evening on day 1 to morning on day 15)
* Cisplatin intravenous administration at a dose of 80 mg/m2 on day 1

ELIGIBILITY:
Inclusion Criteria:

1. Patients with inoperable, locally-advanced or recurrent and/or metastatic gastric adenocarcinoma or gastroesophageal junction adenocarcinoma who are not eligible for curative therapy and are histologically diagnosed.
2. Diseases measurable according to Response Evaluation Criteria in Solid Tumors (RECIST1.1) using imaging technique (CT or MRI).
3. Tissue HER2-negative tumors (primary or metastatic tumors) defined as IHC2+ and FISH- or IHC 0 or 1+ according to gastric cancer assessment system for HER2 (see Annex 12.5).
4. ECOG Performance status 0, 1 or 2 (see Annex 12.1).
5. Survival for at least 3 months should be possible.
6. Appropriate bone marrow, renal, and hepatic functions. General inclusion criteria
7. Males or females aged 19 years.
8. Patients should sign the informed consent form (ICF).

Exclusion Criteria:

1. Patients who previously received chemotherapy for advanced/metastatic diseases (adjuvant/neoadjuvant chemotherapy, completed at least 6 months prior to enrollment in this clinical study, is permitted, but platinum-based adjuvant/neoadjuvant chemotherapy is not permitted).
2. Patients with a lack of physical integration of the upper gastrointestinal tract or with a malabsorption syndrome (e.g., patients who underwent partial or total gastric resection can participate in this clinical study, but patients equipped with a jejunostomy tube cannot participate).
3. Patients with active (serious or uncontrolled) gastrointestinal bleeding.
4. Patients with relevant toxicities remaining following previous curative therapy (except for alopecia). For example, neurotoxicity ≥ grade 2 based on NCI-CTCAE version 5.0.
5. Patients with a history of other malignant diseases based on the date of complete recovery within 5 years prior to the initiation of treatment in this clinical study (except for in-situ cervical cancer and basal cell carcinoma).

   Hematologic, blood chemistry, and organ functions
6. Neutrophil count < 1.5 × 109/L, or platelet count < 100 × 109/L.
7. Serum bilirubin> 1.5 × upper limit of normal (ULN); or AST or ALT > 2.5 × ULN (or > 5 × ULN hepatic metastasis patients); or alkaline phosphatase > 2.5 × ULN (or > 5 × ULN hepatic metastasis patients, or > 10 × ULN hepatic metastasis-free bone metastasis patients); or, albumin < 2.5 g/dL.
8. Creatinine clearance < 60 mL/min. However, creatinine clearance is first calculated using the Cockroft-Gault formula, and if the value is < 60ml/min, a 24hr urine collection test is carried out. Subject enrollment is possible only when creatinine clearance is ≥ 60mL/min.

   Other investigational product-associated exclusion criteria
9. History of proven congestive heart failure; angina pectoris in need of medication; evidence of transmural myocardial infarction through electrocardiogram (ECG); uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg); clinically significant heart valve disorders; and high-risk uncontrolled arrhythmia.
10. Baseline left ventricular ejection fraction (LVEF) < 50% (measured with echocardiogram or MUGA).
11. Patients with dyspnoea at rest due to advanced tumors or other diseases, or who need an adjuvant oxygen therapy.
12. Patients who are treated with long-term or high-dose corticosteroids (steroid inhalation or short-term use of oral steroids for vomiting inhibition and appetite stimulation is permitted).
13. Patients with Clinically significant hypoacusis
14. Patients known to show dihydropyrimidine dehydrogenase (DPD) deficiency. General exclusion criteria
15. Patients with a history of brain metastasis or clinical evidence.
16. Uncontrolled serious systemic intercurrent diseases (e.g., infection or uncontrolled diabetes).
17. Females who are pregnant or are breast-feeding.
18. Fertile males and females who are unwilling to use effective contraceptive methods.
19. Patients who are treated with another investigational product within 4 weeks prior to the initiation of treatment in this clinical study.
20. Patients receiving radiation therapy within 4 weeks prior to the initiation of treatment with the study drug (palliative radiation curative therapy that is partially carried out for bone metastasis. Washout period of 2 weeks is also permitted in patients recovered from all acute toxicities.).
21. Patients who underwent major surgery within 4 weeks prior to the initiation of treatment with the study drug and have not yet been completely recovered.
22. Patients known to have HIV infectivity or active infection with HBV or HCV.
23. Patients with hypersensitivity to the study drug.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Overall tumor response) | 2 years
  Overall tumor response (responder/non-responder) which is a primary efficacy endpoint: is defined as the maximal response among confirmed cases of complete response (CR) or partial response (PR) determined by definite radiological assessment of target and nontarget lesions in accordance with RECIST criteria version 1.1.

SECONDARY OUTCOMES:
progression free survival | 2 years
  Time from the start date of chemotherapy to the date of disease progression or death of any cause which comes first
Duration of response | 2 years
  Time from the date of tumor response by RECIST version 1.1 to the date of disease progression
Overall Survival | 2 years
  Time from the start date of chemotherapy to the date of death of any cause
Time to disease progression | 2 years
  Time from the start date of chemotherapy to the date of disease progression
Safety(Toxicity profile) | 2 years
  Assessed by NCI CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea